CLINICAL TRIAL: NCT04298125
Title: Antenatal Factors Impacting Obesity and Metabolism in Children: Sub-objective 2D
Brief Title: Community Translation of the Expecting Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 260132
Record Dates: First submitted 2020-02-17; First posted 2020-03-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Exercise; Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise in Pregnancy in Community (Experimental): The Expecting intervention at the ACNC includes three 30-45 minute, in-person exercise sessions per week. The sessions are gradually increased in length over the first weeks of participation, and are comprised of 15-30 minutes of moderate aerobic activity (recumbent bike, walking on a treadmill or on an elliptical machine) as well as 5-10 minutes of resistance training using hydraulic exercise equipment. The sessions conclude with stretching exercises. Throughout the session, a personal trainer assesses the rating of perceived exertion using the 6 to 20 point Borg scale of exhaustion.41 Between sessions, participants are asked to monitor their daily step count with a target of 10,000 steps per day using a pedometer provided to the participant. This number is reported to or downloaded by the personal trainer at each in-person session. These elements will be adapted to provide a similar exercise experience that is accessible to women in their local community.
  Interventions: Behavioral: Exercise in Pregnancy
- Standard Care (No Intervention): Participants will receive guidance on exercise from their physician as usual.

INTERVENTIONS:
Behavioral: Exercise in Pregnancy — Women in this group will participate in psychical activity 3 times per week in their community setting.
  Arms: Exercise in Pregnancy in Community

SUMMARY:
The Expecting intervention as delivered in prior studies in a clinical setting is described in a previous approved IRB submission (Protocol 202954). The current project will seek to engage community stakeholders to translate Expecting to a community-delivered intervention and to test its acceptability, feasibility, and fidelity in a proof of principle study with 60 expecting mothers.

DETAILED DESCRIPTION:
The aim of this study is to adapt and determine acceptability, feasibility and fidelity of the research- clinic-based Expecting intervention with pregnant women with obesity in community settings. Specifically, the investigators will show effective application of the Replicating Effective Programs (REP) framework (e.g., fidelity, feasibility, acceptability) to translate the research clinic-based intervention to community settings. REP provides a four-phase process for implementing evidence-based interventions and has demonstrated effective application to translate clinical interventions to community settings. Built into the REP framework is the collection of feedback from community stakeholders, iterative piloting of the intervention in the community, and a process for standardizing the intervention across community settings. Following adaptation, the updated intervention will be piloted. The pilot study will include 60 expecting women. The investigators will randomize half to receive the community-adapted Expecting intervention (Intervention, N=30) and half to receive standard of care (Control, N=30).

ELIGIBILITY:
Inclusion Criteria:

* (a) Body Mass Index > 30,
* (b) singleton pregnancy,
* (c) between 11-15 weeks of pregnancy (at enrollment),
* (d) Do not currently meet recommended guidelines of 150 min of activity per week
* (e) cleared by physician

Exclusion Criteria:

* (a) contraindications for exercise (preeclampsia-eclampsia, premature rupture of the membranes, antepartum hemorrhage, placenta previa, multiple gestation and other defined conditions)
* (b) illicit drug use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This intervention only targets pregnant individuals, which is likely to exclude those who identify as male.
Enrollment: 60 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure:38 weeks | 38 weeks
  Attitudinal Implementation Outcome on a 1 to 5 scale
Acceptability of Intervention Measure: 38 weeks | 38 weeks
  Attitudinal Implementation Outcome on a 1 to 5 scale

SECONDARY OUTCOMES:
Number of intervention sessions completed | 15 weeks through 38 weeks
  Measured with attendance records
Number of minutes of physical activity | Change from Baseline to Delivery and 6 Months Post Delivery
  Measured with Actical
Body Mass Index | Change from Baseline to Delivery and 6 Months Post Delivery
  Collected from Medical Record, weight and height will be combined to report BMI in kg/m^2
Blood Pressure | Change from Baseline to Delivery and 6 Months Post Delivery
  Collected from Medical Record
Total Cholesterol from Lipid Panel | Change from Baseline to Delivery and 6 Months Post Delivery
  Collected from Medical Record

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swindle T, Martinez A, Borsheim E, Andres A. Adaptation of an exercise intervention for pregnant women to community-based delivery: a study protocol. BMJ Open. 2020 Sep 6;10(9):e038582. doi: 10.1136/bmjopen-2020-038582. PMID 32895286

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04298125/Prot_SAP_000.pdf